CLINICAL TRIAL: NCT04397224
Title: Prospective Multicenter Observation Study on the Serial Changes in Ventriculo-ventricular Conduction Times According to Cardiac-resynchronization Therapy Response
Brief Title: Reduction or Extension of COnduction Time With Ventricular Electromechanical Remodeling (RECOVER)
Acronym: RECOVER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-05-073
Record Dates: First submitted 2020-05-17; First posted 2020-05-21 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CRT responder
  Interventions: Diagnostic Test: Device interrogation
- CRT non-responder
  Interventions: Diagnostic Test: Device interrogation

INTERVENTIONS:
Diagnostic Test: Device interrogation — Ventriculo-ventricular conduction time measurement using device analyzer

SUMMARY:
This prospective multicenter registry study aims to detect the serial changes in ventriculo-ventricular conduction times according to cardiac-resynchronization therapy response.

ELIGIBILITY:
Inclusion Criteria:

* meeting the current ESC or ACCF/AHA/HRS Class I or Class IIa indications for cardiac-resynchronization (CRT) implant

Exclusion Criteria:

* Myocardial infarction, unstable angina within 40 days prior the enrollment
* Recent cardiac revascularization in the 4 weeks prior to the enrollment or planned for the 3 months following
* Cerebrovascular accident (CVA) or transient ischemic attack (TIA) in the 3 months prior to the enrollment
* Primary valvular disease requiring surgical correction
* Pregnant or are planning during the duration of the investigation
* Status 1 candidate for cardiac transplantation or consideration for transplantation over the next 12 months
* Post-cardiac transplantation
* Life expectancy < 12 months
* Currently participating in any other clinical investigation except for observational registry

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients implanted with multipoint pacing CRT device and quadripolar left ventricular lead from Abbott
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-07-20 (Actual); Primary Completion 2022-07-20 (Estimated); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
Serial change of ventriculo-ventricular conduction times | from enrollment to last follow-up (2 years)
  Reduction or extension of ventriculo-ventricular conduction times

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - Sejong General Hospital, Bucheon-si
  - Samsung Changwon Medical Center, Changwon
  - Chungnam National University Hospital, Daejeon
  - Eulji University Hospital, Daejeon
  - Seoul National University Bundang Hospital, Seongnam
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided